CLINICAL TRIAL: NCT05942131
Title: The Effect of Group-Based Laughter Yoga on the Level of Secondary Traumatic Stress and Depression Experienced by Midwifery Students After the Earthquake
Brief Title: The Effect of Group-Based Laughter Yoga on Midwifery Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Assoc. Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBÜ-AYDINKARTAL-005
Record Dates: First submitted 2023-06-24; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Laughter Yoga
Keywords: secondary trauma; depression; midwifery student; earthquake
MeSH Terms: conditions — Compassion Fatigue; Depression

STUDY DESIGN:
Intervention Model Description: Single blind randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (n:42) (Experimental): Laughter yoga will be practiced to students in the intervention group
  Interventions: Other: Group-based laughter yoga
- Control Group (n:42) (No Intervention): No intervention will be applied to the control group midwives and "Secondary Traumatic Stress Scale for Social Media Users" and "Beck Depression Inventory" will be applied when they are included in the study and again after 4-6 weeks.

INTERVENTIONS:
Other: Group-based laughter yoga — A total of 8 sessions of laughter yoga will be applied to the students in the intervention group, 2 sessions per week. Each session will last 45 minutes on average. Each session will consist of groups of 7 people. An information meeting about the sessions will be held with the midwifery students who volunteered to participate in the study and assigned to the intervention group before starting laughter yoga. Midwifery students will be administered "Secondary Traumatic Stress Scale for Social Media Users" and "Beck Depression Inventory" before and after 4-6 weeks.
  Arms: Intervention Group (n:42)

SUMMARY:
This study was planned to determine the effect of laughter yoga on the secondary traumatic stress and depression levels experienced by midwifery students due to the use of social media after the earthquake. The universe of the research will be the third year students of Health Sciences University Hamidiye Health Sciences Faculty Midwifery Department (N:84).

A total of 8 sessions of laughter yoga, 2 sessions per week, will be applied to midwifery students in the intervention group of the research. It will be determined as intervention (n:42) and control (n:42) groups. "Descriptive Information Form", "Secondary Traumatic Stress Scale for Social Media Users" and "Beck Depression Inventory" will be applied to both groups.

DETAILED DESCRIPTION:
It was planned to determine the effect of laughter yoga on the secondary traumatic stress and depression levels experienced by midwifery students due to the use of social media after the earthquake. The study will be implemented according to the CONSORT 2010 guidelines.

The research will be carried out in Health Sciences University, Hamidiye Faculty of Health Sciences, Midwifery department classroom. In pre-research classrooms; An environment with good lighting, sound systems and allowing individuals to move comfortably will be arranged. Hamidiye Faculty of Health Sciences Midwifery Department 3rd year students who volunteered to participate in the study will be determined as the intervention (n:42) and control (n:42) groups with the numbers assigned by the researchers via the https://www.randomizer.org/ site. An introductory information form will be applied to all students. A total of 8 sessions of laughter yoga, 2 sessions per week, will be applied to midwifery students in the intervention group of the research. Laughter yoga will be practiced by researchers with leadership certification. Each session will take an average of 45 minutes. Each session will consist of groups of 7 people. Before starting the laughter yoga session, an information meeting will be held with midwifery students who volunteered to participate in the study and were assigned to the intervention group. Midwifery students will be administered "Secondary Traumatic Stress Scale for Social Media Users" and "Beck Depression Inventory" before and 4-6 weeks after the application. No intervention will be applied to the control group midwives, and "Secondary Traumatic Stress Scale for Social Media Users" and "Beck Depression Inventory" will be administered again when they are included in the study and 4-6 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Being an active student in the 3rd year of Health Sciences University, Hamidiye Faculty of Health Sciences, Department of Midwifery
* Volunteering to participate in research

Exclusion Criteria:

* Having a psychiatric diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | 1 hour before laughter yoga practice
  In this form, which was created by the researchers based on the literature, participants' age, high school they graduated from, secondary traumatic stress experience, etc. questions are included.
Beck Depression Inventory (BDI) | 1 hour before laughter yoga practice
  The scale designed to determine the depressive levels of individuals consists of 21 items. The aim of the inventory is not to diagnose depression but to express the degree of depressive symptoms numerically. Higher scores indicate an increase in depressive symptoms. Each item receives a score between 0-3 and the scores that can be obtained from the inventory are between 0-63. The scores of 0-9 points indicate normal, 10-18 points indicate mild, 19-29 points indicate moderate, and 30-63 points indicate severe depressive symptoms.
Secondary Traumatic Stress Scale for Social Media Users | 1 hour before laughter yoga practice
  The scale was developed to examine avoidance and arousal symptoms associated with indirect exposure to traumatic experiences through social media users. The scale consists of 17 items. The scale was reduced to a single-factor structure. There are no reverse coded items. The lowest score that can be obtained from the scale is 17 and the highest score is 85. As the total score obtained from the scale increases, individuals' secondary traumatic stress caused by social media increases.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | 4-6 weeks after application
  The scale designed to determine the depressive levels of individuals consists of 21 items. The aim of the inventory is not to diagnose depression but to express the degree of depressive symptoms numerically. Higher scores indicate an increase in depressive symptoms. Each item receives a score between 0-3 and the scores that can be obtained from the inventory are between 0-63. The scores of 0-9 points indicate normal, 10-18 points indicate mild, 19-29 points indicate moderate, and 30-63 points indicate severe depressive symptoms.
Secondary Traumatic Stress Scale for Social Media Users | 4-6 weeks after application
  The scale was developed to examine avoidance and arousal symptoms associated with indirect exposure to traumatic experiences through social media users. The scale consists of 17 items. The scale was reduced to a single-factor structure. There are no reverse coded items. The lowest score that can be obtained from the scale is 17 and the highest score is 85. As the total score obtained from the scale increases, individuals' secondary traumatic stress caused by social media increases.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No